CLINICAL TRIAL: NCT06895525
Title: The HEART Study: A Randomized, Double-Blind, Parallel Placebo-Controlled Trial on the Efficacy of HellenCare in Early-Stage Alzheimer's Disease
Brief Title: Efficacy of HellenCare in Early-Stage Alzheimer's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBJ-01
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer's Disease Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HellenCare (Experimental)
  Interventions: Dietary Supplement: HellenCare
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: HellenCare — 2 g, twice daily, to be taken on an empty stomach.
  Arms: HellenCare
Dietary Supplement: Placebo — 2 g, twice daily, to be taken on an empty stomach.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate whether HellenCare, a multicomponent nutraceutical, improves cognitive and functional outcomes in patients with early-stage Alzheimer's disease (AD). The investigators will compare changes in outcomes between the HellenCare group and the placebo group to determine if the intervention is effective and safe.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 50 to 85 years
* Clinically diagnosed for the first time with probable Alzheimer's disease dementia (AD dementia) or AD-related mild cognitive impairment (MCI) according to the National Institute on Aging-Alzheimer's Association (NIA-AA) core clinical criteria.
* MMSE (Mini-Mental State Examination): Score between 22 and 30.
* CDR (Clinical Dementia Rating): Total score of 0.5 or 1. Memory domain score on CDR: ≥0.5.
* Able to comply with study procedures and attend scheduled visits.
* Willingness to participate and provide informed consent.

Exclusion Criteria:

* Presence of other dementia-causing conditions (e.g., vascular dementia, Lewy body dementia, etc)
* Severe neurological comorbidities (e.g., history of seizures, cerebral infarction, intracerebral hemorrhage, traumatic brain injury, brain tumors, etc.)
* Presence of severe anxiety, depression, schizophrenia, bipolar disorder, or other psychotic disorders requiring active treatment.
* History of alcohol or drug dependence within the past 1 year.
* Allergies to study dietary supplement.
* Use of anti-dementia medications ( e.g., donepezil, galantamine, memantine, etc).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Clinical Dementia Rating-Sum of Boxes (CDR-SB) from baseline | Baseline to three months
  CDR-SB range 0-18, with higher scores indicating more severe dementia.

SECONDARY OUTCOMES:
Changes in Mini-Mental State Examination (MMSE) Scores from Baseline | Up to Day 90 (including baseline and follow-up visits).
  MMSE range 0-30, with higher scores indicating better cognitive functioning.
Changes in Montreal Cognitive Assessment (MoCA) Scores from Baseline | Up to Day 90 (including baseline and follow-up visits).
  MoCA range 0-30, with higher scores indicating better cognitive functioning.
Changes in Neuropsychiatric Inventory (NPI) from Baseline | Up to Day 90 (including baseline and follow-up visits).
  NPI score range is 0-144 for patient assessment and 0-60 for caregiver distress assessment. In patient assessment, higher scores indicate more severe neuropsychiatric disorders; in caregiver distress assessment, higher scores indicate greater distress.
Changes in Alzheimer's Disease Cooperative Study-Activities of Daily Living（ADCS-ADL）from baseline | Up to Day 90 (including baseline and follow-up visits).
  ADCS-ADL range 0-78, with higher scores indicating better functional ability in daily activities.
Changes in Geriatric Depression Scale (GDS) from Baseline | Up to Day 90 (including baseline and follow-up visits).
  GDS is a standardized assessment tool for evaluating depressive symptoms in older adults, scored from 0 to 15, with higher scores indicating greater severity of depressive symptoms and associated functional impairment.
Changes in Self-Rating Anxiety Scale (SAS) from Baseline | Up to Day 90 (including baseline and follow-up visits).
  The SAS has a range of 20-80, with higher scores indicating more severe anxiety symptoms.
Changes in Self-Rating Depression Scale (SDS) from Baseline | Up to Day 90 (including baseline and follow-up visits).
  The SDS has a range of 20-80, with higher scores indicating more severe depressive symptoms.
Changes in Self-Rating Scale of Sleep (SRSS) from Baseline | Up to Day 90 (including baseline and follow-up visits).
  The SRSS has a range of 10-50, with higher scores indicating more severe sleep problems.
Changes in plasma biomarker levels from baseline | Baseline to three months
  The plasma biomarkers include Aβ42/40，p-tau181, p-tau217, NfL and GFAP
Safety and Tolerability | Up to Day 90 (including baseline and follow-up visits).
  The adverse event, discontinuation due to intolerability, etc will be monitored.